CLINICAL TRIAL: NCT01381133
Title: Adolescent Outpatient and Continuing Care Study
Acronym: AOCCS
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Chestnut Health Systems (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Treatment
Other Study IDs: 1022-0602; R01DA018183 (NIH); U79TI13356 (Other Grant/Funding Number: DHHS)
Record Dates: First submitted 2011-06-23; First posted 2011-06-27 (Estimated); Last update posted 2013-08-14 (Estimated); Status verified 2013-08

CONDITIONS: Substance Abuse; Substance Dependence
Keywords: Substance abuse; Adolescent outpatient treatment; Continuing care; Outcomes
MeSH Terms: conditions — Substance-Related Disorders | interventions — Motivational Interviewing

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- CBOP without ACC (Experimental)
  Interventions: Behavioral: Chestnut Bloomington Outpatient (CBOP)
- CBOP with ACC (Experimental)
  Interventions: Behavioral: Chestnut Bloomington Outpatient (CBOP); Behavioral: Assertive Continuing Care (ACC)
- MET/CBT 7 without ACC (Experimental)
  Interventions: Behavioral: Motivational Enhancement Therapy/Cognitive Behavior Treatment (MET/CBT 7)
- MET/CBT 7 with ACC (Experimental)
  Interventions: Behavioral: Motivational Enhancement Therapy/Cognitive Behavior Treatment (MET/CBT 7); Behavioral: Assertive Continuing Care (ACC)

INTERVENTIONS:
Behavioral: Chestnut Bloomington Outpatient (CBOP) — CBOP is an evidence-informed intervention that has developed over 20 years and been shaped by treatment research. The underlying theory of change is that the combination of multiple evidence-based and best-practice treatment components will increase the adolescent's desire to change, provide the necessary skills, and create an environment supportive for this change. The intervention is based on a manual and is primarily delivered through skill and therapy groups, combined with a limited number of family and individual sessions for treatment planning and progress reviews.
  Arms: CBOP with ACC; CBOP without ACC
Behavioral: Motivational Enhancement Therapy/Cognitive Behavior Treatment (MET/CBT 7) — A manual-based 5-session MET/CBT model was supplemented with 2 family sessions. First was a family session to provide parents with an overview. Next was an individual adolescent MET session that focused on building rapport, explaining treatment, building motivation, and reviewing personalized feedback. In the third session, the therapist helped the adolescent complete a functional analysis of substance use and a personal goal worksheet. During sessions 4-6, the adolescent joined a closed group of 6 for 90-min CBT skills groups focusing on substance refusal skills, enhancing social support, planning for high-risk situations, and coping with relapse. The last session was a family session to review progress, relapse signs, and continuing care plans. Treatment lasted about 12 weeks.
  Arms: MET/CBT 7 with ACC; MET/CBT 7 without ACC
Behavioral: Assertive Continuing Care (ACC) — ACC is a home-based continuing care approach that takes place over a 12-14 week period and has shown promise in a randomized clinical trial of adolescents discharged from residential treatment. Following an operant reinforcement and skills training model, ACC combines the Adolescent Community Reinforcement Approach and case management services to help adolescents and their caregivers engage in prosocial activities, skills, and needed community services during weekly home visits.
  Arms: CBOP with ACC; MET/CBT 7 with ACC

SUMMARY:
The purpose of this study was to evaluate the effectiveness and cost-effectiveness of two types of outpatient treatment with and without Assertive Continuing Care (ACC) for 320 adolescents with substance use disorders. Study participants were randomly assigned to one of four conditions: (a) Chestnut's Bloomington Outpatient Treatment (CBOP) without ACC; (b) CBOP with ACC; (c) Motivational Enhancement Therapy/Cognitive Behavior Therapy-7 session model (MET/CBT7) without ACC; and (d) MET/CBT7 with ACC. Based on prior quasi and experimental studies, the investigators hypothesized that MET/CBT would be more effective and cost-effective than CBOP in terms of increasing days abstinent and decreasing substance abuse problems. Additionally, the investigators hypothesized that the groups receiving ACC would have significantly better outcomes than the groups without ACC. Lastly, the investigators hypothesized that adding ACC to MET/CBT would be the most cost-effective option in terms of days abstinent.

DETAILED DESCRIPTION:
This study evaluated the effectiveness and cost-effectiveness of two types of outpatient treatment with and without Assertive Continuing Care (ACC) for 320 adolescents with substance use disorders. Study participants were randomly assigned to one of four conditions: (a) Chestnut's Bloomington Outpatient Treatment (CBOP) without ACC; (b) CBOP with ACC; (c) Motivational Enhancement Therapy/Cognitive Behavior Therapy-7 session model (MET/CBT7) without ACC; and (d) MET/CBT7 with ACC. All study conditions attained high rates of participant engagement and retention. Follow-up interviews were completed with over 90% of the adolescents at three, six, nine, and 12 months after treatment admission. There was a significant time by condition effect over 12 months, with CBOP having a slight advantage for average percentage of days abstinent. Unlike previous findings that ACC provided incremental effectiveness following residential treatment, there were no statistically significant findings with regard to the incremental effectiveness of ACC following outpatient treatment. Analysis of the costs of each intervention combined with its outcomes revealed that the most cost-effective condition was MET/CBT7 without ACC.

ELIGIBILITY:
Inclusion Criteria:

* 12-18 years old
* met ASAM's (2001) Patient Placement Criteria for Level I outpatient treatment based on a substance abuse or dependence diagnosis and six dimensional admission criteria (i.e., severity of intoxication/withdrawal, physical health, emotional/behavioral health, treatment readiness, relapse potential, and recovery environment)
* attended an admission appointment

Exclusion Criteria:

* "stepped-down" from residential treatment and were therefore more severe than adolescents who entered outpatient treatment from the community
* were recommended only for individual counseling, as both outpatient treatment conditions had group components
* were a ward of the state
* did not have a parent/guardian present during admission to outpatient treatment
* appeared to have insufficient mental capacity to provide informed consent
* did not speak English with sufficient ability to understand study procedures and instruments

Ages: 12 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 320 (Actual)
Dates: Start 2002-09; Primary Completion 2008-12 (Actual); Study Completion 2008-12 (Actual)

PRIMARY OUTCOMES:
Change in Percentage of days abstinent from any alcohol and drugs | Baseline and 3, 6, 9, and 12 months post-baseline
Change in Days abstinent from alcohol alone | Baseline and 3, 6, 9, and 12 months post-baseline
Change in Substance use problems | Baseline and 3, 6, 9, and 12 months post-baseline
  Measured using the Substance Problem Scale of the Global Appraisal of Individual Needs
Change in Recovery status | 12 months post-baseline
  Being in recovery at the end of the study was defined as living in the community (vs. being incarcerated, or residing in inpatient treatment or other controlled environment) and reporting no past month substance use, abuse, or dependence problems at the 12 month interview. Urine samples were collected as described above in Section 2.4.2, and when an adolescent reported being in recovery but the urine test result suggested a false-negative self-report, data were re-coded to show the adolescent as not being in recovery.

CONTACTS AND LOCATIONS:
Overall Officials: Susan H Godley, Ph.D., Principal Investigator — Chestnut Health Systems
Locations (1):
- Chestnut Health Systems, Bloomington, Illinois, United States

REFERENCES:
- [Result] Godley SH, Garner BR, Passetti LL, Funk RR, Dennis ML, Godley MD. Adolescent outpatient treatment and continuing care: main findings from a randomized clinical trial. Drug Alcohol Depend. 2010 Jul 1;110(1-2):44-54. doi: 10.1016/j.drugalcdep.2010.02.003. Epub 2010 Mar 9. PMID 20219293
- See also: MET/CBT 5 manual — http://www.chestnut.org/Portals/14/PDF_Documents/Lighthouse/CYT/Products/MCB5_CYT_v1.pdf
- See also: ACC: A-CRA manual (used in conjunction with case management manual) — http://www.chestnut.org/Portals/14/PDF_Documents/Lighthouse/CYT/Products/ACRA_CYT_v4.pdf
- See also: ACC: case management manual (used in conjunction with A-CRA manual) — http://www.chestnut.org/Portals/14/PDF_Documents/Lighthouse/Manuals/ACC_manual_revised_2nd_ed_111306.pdf